CLINICAL TRIAL: NCT04201496
Title: SGLT2 Inhibitor Adjunctive Therapy to Closed Loop Control in Type 1 Diabetes Mellitus
Acronym: CiQ-SGLT2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ananda Basu, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ananda Basu, MD, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 190017; DP3DK106785 (NIH)
Record Dates: First submitted 2019-11-04; First posted 2019-12-17 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes
Keywords: Artificial Pancreas (AP); Sodium-glucose co-transporter 2 (SGLT2) inhibitor; Insulin Pumps; Continuous Glucose Monitor (CGM); Closed Loop Control; Low blood glucose index (LBGI); High blood glucose index (HBGI)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Participants will be first randomized to taking empagliflozin or not taking this drug. Participants will then be randomized to using the Basal-IQ insulin pump first or the Control-IQ insulin pump first. Participants then transition to using the other pump.
  With empagliflozin:
  * Control-IQ x 4 weeks (CiQ-EMPA) then Basal-IQ x 2 weeks (BiQ-EMPA)
  * Basal-IQ x 2 weeks (BiQ-EMPA) then Control-IQ x 4 weeks (CiQ-EMPA)
  Without empagliflozin:
  * Control-IQ x 4 weeks (CiQ-NO EMPA) then Basal-IQ x 2 weeks (BiQ-NO EMPA)
  * Basal-IQ x 2 weeks (BiQ-NO EMPA) then Control-IQ x 4 weeks (CiQ-NO EMPA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Empagliflozin + Control-IQ x 4 wks then Basal-IQ x 2 wks (Experimental): Control-IQ x 4 weeks (CiQ-EMPA) then Basal-IQ x 2 weeks (BiQ-EMPA)
  Interventions: Combination Product: Empagliflozin + Control-IQ x 4 wks then Basal-IQ x 2 wks
- Empagliflozin + Basal-IQ x 2 wks then CiQ x 4 wks (Experimental): Basal-IQ x 2 weeks (BiQ-EMPA) then Control-IQ x 4 weeks (CiQ-EMPA)
  Interventions: Combination Product: Empagliflozin + Basal-IQ x 2 wks then Control-IQ x 4 wks
- No Empagliflozin + Control-IQ x 4 wks then Basal-IQ x 2 wks (Active Comparator): Control-IQ x 4 weeks (CiQ-NO EMPA) then Basal-IQ x 2 weeks (BiQ-NO EMPA)
  Interventions: Device: No Empagliflozin + Control-IQ x 4 wks then Basal-IQ x 2 wks
- No Empagliflozin + Basal-IQ x 2 wks then Control-IQ x 4 wks (Active Comparator): Basal-IQ x 2 weeks (BiQ-NO EMPA) then Control-IQ x 4 weeks (CiQ-NO EMPA)
  Interventions: Device: No Empagliflozin + Basal-IQ x 2 wks then Control-IQ x 4 wks

INTERVENTIONS:
Combination Product: Empagliflozin + Control-IQ x 4 wks then Basal-IQ x 2 wks — Participants with be provided with Empagliflozin to take daily for approximately 10 weeks. Along with the study medication, participants will initially use the Tandem t:slim insulin pump with Control-IQ Technology for 4 weeks. Participants will then transition to using the Tandem t:slim insulin pump with Basal-IQ Technology for 2 weeks.
  Arms: Empagliflozin + Control-IQ x 4 wks then Basal-IQ x 2 wks
Combination Product: Empagliflozin + Basal-IQ x 2 wks then Control-IQ x 4 wks — Participants with be provided with Empagliflozin to take daily for approximately 10 weeks. Along with the study medication, participants will initially use the Tandem t:slim insulin pump with Basal-IQ Technology for 2 weeks. Participants will then transition to using the Tandem t:slim insulin pump with Control-IQ Technology for 4 weeks.
  Arms: Empagliflozin + Basal-IQ x 2 wks then CiQ x 4 wks
Device: No Empagliflozin + Control-IQ x 4 wks then Basal-IQ x 2 wks — Participants will initially use the Tandem t:slim insulin pump with Control-IQ Technology for 4 weeks. Participants will then transition to using the Tandem t:slim insulin pump with Basal-IQ Technology for 2 weeks. Empaglizflozin will not be provided to this group.
  Arms: No Empagliflozin + Control-IQ x 4 wks then Basal-IQ x 2 wks
Device: No Empagliflozin + Basal-IQ x 2 wks then Control-IQ x 4 wks — Participants will initially use the Tandem t:slim insulin pump with Basal-IQ Technology for 2 weeks. Participants will then transition to using the Tandem t:slim insulin pump with Control-IQ Technology for 4 weeks. Empaglizflozin will not be provided to this group.
  Arms: No Empagliflozin + Basal-IQ x 2 wks then Control-IQ x 4 wks

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of combining SGLT2 inhibitors with closed loop control (CLC).

DETAILED DESCRIPTION:
The first five participants will be enrolled in a Pilot Study to use the Basal-IQ with Empagliflozin 10 mg daily for approximately two weeks. These participants will participate in an estimated 36-48-hour hotel admission to initiate use of Closed Loop Control. The safety data from the Pilot Study will be presented to the Data Safety Monitoring Board (DSMB) for review.

Upon DSMB approval, approximately 40 participants will be randomized 1:1 in a crossover design. Participants will use empagliflozin 5 mg daily. This main study is a randomized control trial where approximately 50 participants, aged 18 to less than 65 y.o. at time of consent, will be in the trial for up to 10 weeks.

With empagliflozin:

* Control-IQ (CiQ) x 4 weeks (CiQ-EMPA) then Basal-IQ x 2 weeks (BiQ-EMPA)
* Basal-IQ x 2 weeks (BiQ-EMPA) then CiQ x 4 weeks (CiQ-EMPA)

Without empagliflozin:

* CiQ x 4 weeks (CiQ-NO EMPA) then Basal-IQ x 2 weeks (BiQ-NO EMPA)
* Basal-IQ x 2 weeks (BiQ-NO EMPA) then CiQ x 4 weeks (CiQ-NO EMPA)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 and ≤65 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
3. Currently using an insulin pump for at least six months
4. Currently using insulin for at least six months
5. Using insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
6. Access to internet and willingness to upload data during the study as needed
7. For females, not currently known to be pregnant or breastfeeding
8. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
9. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use
10. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study
11. Total daily insulin dose (TDD) at least 10 U/day
12. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, biguanides, sulfonylureas and naturaceuticals)
13. Willingness to eat at least 100 grams of carbohydrates per day
14. An understanding and willingness to follow the protocol and signed informed consent
15. Pilot Participants: Agree to hotel/research house admission with other Pilot participants on a date selected by the study team.

Exclusion Criteria:

1. Hemoglobin A1c >9%
2. History of diabetic ketoacidosis (DKA) in the 12 months prior to enrollment
3. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
4. Pregnancy or intent to become pregnant during the trial
5. Currently breastfeeding or planning to breastfeed
6. Currently being treated for a seizure disorder
7. Planned surgery during study duration
8. History of cardiac arrhythmia (except for benign premature atrial contractions and benign premature ventricular contractions which are permitted)
9. Clinically significant electrocardiogram (ECG) abnormality at time of Screening, as interpreted by the study medical physician
10. Use of diuretics (e.g. Lasix, Thiazides)
11. History of chronic or recurrent genital infections
12. eGFR lab value below 60 mL/min/1.73 m2
13. Treatment with any non-insulin glucose-lowering agent (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals)
14. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

    1. Severe renal impairment, end-stage renal disease, or dialysis
    2. Inpatient psychiatric treatment in the past six months
    3. Presence of a known adrenal disorder
    4. Abnormal liver function test results (Transaminase>2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
    5. Uncontrolled thyroid disease
15. Severe renal impairment, end-stage renal disease, or dialysis
16. Use of an automated insulin delivery mechanism that is not downloadable by the subject or study team
17. Current enrollment in another clinical trial, unless approved by the investigator of both studies or if clinical trial is a non-interventional registry trial
18. Alcohol restricted to no more than 2 drinks per night in men and no more than 1 drink per night in women
19. Low carb diet (less than 100g per day)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
CGM-measured time in the target range 70-180mg/dl (TIR) during the day | 6 weeks
  CGM-measured time in the target range 70-180mg/dl (TIR) during the day

SECONDARY OUTCOMES:
Time below 70 mg/dl | 6 weeks
  Time below 70 mg/dl
Time above 180 mg/dl | 6 weeks
  Time above 180 mg/dl
Time between 70-140 mg/dl 5 hours post prandial | 6 weeks
  Time between 70-140 mg/dl 5 hours post prandial
Glucose variability index HBGI | 6 weeks
  Glucose variability index HBGI
Glucose variability index LBGI | 6 weeks
  Glucose variability index LBGI
Glucose variability index ADRR | 6 weeks
  Glucose variability index ADRR
Safety evaluation of empagliflozin as adjuvant therapy added to a closed loop artificial pancreas system | 6 weeks
  Number of episodes of diabetic ketoacidosis (DKA)
Safety evaluation of empagliflozin as adjuvant therapy added to a closed loop artificial pancreas system | 6 weeks
  Number of episodes of severe hypoglycemia (glucose <50 mg/dl)
Episodes of diabetes ketoacidosis (DKA) | 6 weeks
  The number of DKA events in the experimental group as compared to the control group
Episodes of severe hypoglycemia (glucose <50 mg/dL) | 6 weeks
  The number of hypoglycemic events in the experimental group as compared to the control group
Genital infections | 6 weeks
  Number of genital infections (balanitis, urethritis, vulvar infections, Fournier's gangrene) that occur in the experimental group versus the control group
Urinary Tract Infections | 6 weeks
  Number of urinary tract infections that occur in the experimental group versus the control group
Total amount of insulin used | 6 weeks
  The number of amount of insulin used in the experimental group as compared to the control group
Number of hyperglycemic episodes as defined by contiguous CGM above 300 mg/dL | 6 weeks
  Number of hyperglycemic episodes, defined as contiguous CGM values above 300 mg/dL, that occur in the experimental group versus the control group

CONTACTS AND LOCATIONS:
Overall Officials: Ananda Basu, MD, Principal Investigator — University of Virginia; Ralf Nass, MD, Study Chair — University of Virginia
Locations (1):
- University of Virginia, Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
To be determined
Supporting Information: Study Protocol
Time Frame: After publication for one year

REFERENCES:
- [Derived] Garcia-Tirado J, Farhy L, Nass R, Kollar L, Clancy-Oliveri M, Basu R, Kovatchev B, Basu A. Automated Insulin Delivery with SGLT2i Combination Therapy in Type 1 Diabetes. Diabetes Technol Ther. 2022 Jul;24(7):461-470. doi: 10.1089/dia.2021.0542. Epub 2022 Mar 14. PMID 35255229

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT04201496/Prot_SAP_002.pdf
  • Informed Consent Form (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT04201496/ICF_003.pdf